CLINICAL TRIAL: NCT00695890
Title: Effects of Sevoflurane and Propofol on Light Flash Evoked Pupillometry.
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 012007070222
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Measurement of Pupil Diameter
Keywords: Pupillometry; Sevoflorane; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy volunteers

SUMMARY:
Null hypothesis (HO): There will be no difference in pupillometry readings when using any of the maintenance anesthetic techniques within subjects.

Alternate hypothesis (HA): Pupillometry readings will be affected by a change in the anesthetic technique

DETAILED DESCRIPTION:
Postoperative visual loss resulting from a surgical procedure not performed on the eye is a devastating outcome for the patient and poorly understood by the medical community. It is potentially a preventable complication. Diminished blood supply to the optic nerve, affecting both the anterior or posterior portions of the optic nerve, is the most common cause of postoperative visual loss. Other, less common causes include occlusion of the retinal artery and vein, a retinal embolism and cortical blindness. The incidence of postoperative visual loss increases in patients undergoing cardiopulmonary bypass and prone spine surgery. Although the etiology of post-operative visual loss is unknown, it is thought to be multifactorial, and several potential risk factors have been identified, including degree of low blood pressure, preoperative hematocrit, external compression of the eye, amount of blood loss, prolonged duration of surgical time and increased pressure in the eye associated with positioning. To date studies have focused on the mechanism associated with the visual loss. We would like to focus on the feasibility of using a monitor which may signal loss of visual function intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70 years of age who are mentally capable of providing an informed consent and who are medically classified as ASA 1 or 2.
* Planned elective orthopedic extremity surgery in the supine position with the head in the neutral position.

Exclusion Criteria:

* Failure to provide an informed consent
* Known history of eye disease which cannot be corrected with lenses
* Surgery lasting less than 45 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
We would like to focus on the feasibility of using a monitor which may signal loss of visual function intraoperatively. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Geordie Grant, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ, Newark, New Jersey, United States